CLINICAL TRIAL: NCT06459401
Title: Effects of an Overground Propulsion Neuroprosthesis in Community-dwelling Individuals After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Harvard University (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); American Heart Association (Other)
Responsible Party: Principal Investigator, Lou Awad, PT, DPT, PhD, Professor, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5715; 830019 (Other Grant/Funding Number: American Heart Association Pre-Doctoral Fellowship Award); U54EB015408 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-06-14 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: Gait Rehabilitation; Functional Electrical Stimulation (FES); Stroke; Exosuit; Propulsion; Neuroprosthesis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: All participants with stroke will complete study procedures that include walking with and without the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Neuroprosthesis-Assisted Walking Evaluation (Experimental): Participants with chronic stroke will perform a series of short overground walking evaluations at a self-selected fast walking speed with the neuroprosthesis powered and unpowered. When the neuroprosthesis is powered, it provides active neurostimulation assistance for foot clearance and propulsion. When the neuroprosthesis is unpowered, it is worn by the participant but does not provide active assistance.
  Interventions: Device: Propulsion Neuroprosthesis

INTERVENTIONS:
Device: Propulsion Neuroprosthesis — A neuroprosthesis is a textile-based surface neurostimulation system worn on the waist and paretic lower limb that delivers neurostimulation assistance via electroconductive pads placed on the skin over the target muscles. The neuroprosthesis provides dorsiflexor stimulation during swing phase for foot clearance and plantarflexor stimulation during stance phase for propulsion, delivered synchronously based on integrated sensors detecting the wearer's gait pattern.

SUMMARY:
This interventional study evaluates the effects of an overground propulsion neuroprosthesis that delivers adaptive neurostimulation assistance to the paretic plantarflexors and dorsiflexors of people post-stroke. Individuals with chronic post-stroke hemiparesis will walk with and without the neuroprosthesis overground and on a treadmill. The goal of the study is to understand how adaptive neurostimulation delivered by the neuroprosthesis affects clinical and biomechanical measures of walking function in order to guide future rehabilitation approaches for restoring walking ability after stroke.

DETAILED DESCRIPTION:
This interventional study evaluates the effects of an overground propulsion neuroprosthesis that delivers adaptive neurostimulation assistance to the paretic plantarflexors and dorsiflexors of people post-stroke. Individuals with chronic post-stroke hemiparesis will walk with and without the neuroprosthesis overground and on a treadmill. The goal of the study is to understand how adaptive neurostimulation delivered by the neuroprosthesis affects clinical and biomechanical measures of walking function in order to guide future rehabilitation approaches for restoring walking ability after stroke.

Ten individuals with chronic post-stroke hemiparesis will complete a single session of walking with and without the neuroprosthesis. Study evaluations will be conducted both before and after the session, without the neuroprosthesis active, and during the neuroprosthesis-supported walking.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a stroke event occurring at least 6 months ago
* Observable gait deficits
* Independent ambulation for at least 30 meters (using an assistive device as needed but without a rigid brace or ankle foot orthosis)
* Passive ankle dorsiflexion range of motion to neutral with the knee extended
* Ability to follow a 3-step command
* Resting heart rate between 40-100 bpm
* Resting blood pressure between 90/60 and 170/90 mmHg
* NIH Stroke Scale Question 1b score > 1 and Question 1c score > 0
* HIPAA Authorization to allow communication with healthcare provider
* Medical clearance by a physician

Exclusion Criteria:

* Severe aphasia or inability to communicate with investigators
* Neglect or hemianopia
* Serious comorbidities that may interfere with ability to participate in the research (e.g. musculoskeletal, cardiovascular, pulmonary)
* Pacemakers or similar electrical implants that could be affected by electrical stimulation
* Metal implants directly under the stimulation sites
* Pressure ulcers or skin wounds located near human-device interface sites
* More than 2 unexplained falls in the previous month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Awad, PT, DPT, PhD, Study Director — Boston University
Locations (2):
- United States (2):
  - Science and Engineering Complex, Boston, Massachusetts
  - Neuromotor Recovery Laboratory, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awad LN, Kesar TM, Reisman D, Binder-Macleod SA. Effects of repeated treadmill testing and electrical stimulation on post-stroke gait kinematics. Gait Posture. 2013 Jan;37(1):67-71. doi: 10.1016/j.gaitpost.2012.06.001. Epub 2012 Jul 15. PMID 22796242
- [Background] Kesar TM, Perumal R, Jancosko A, Reisman DS, Rudolph KS, Higginson JS, Binder-Macleod SA. Novel patterns of functional electrical stimulation have an immediate effect on dorsiflexor muscle function during gait for people poststroke. Phys Ther. 2010 Jan;90(1):55-66. doi: 10.2522/ptj.20090140. Epub 2009 Nov 19. PMID 19926681
- [Background] Hakansson NA, Kesar T, Reisman D, Binder-Macleod S, Higginson JS. Effects of fast functional electrical stimulation gait training on mechanical recovery in poststroke gait. Artif Organs. 2011 Mar;35(3):217-20. doi: 10.1111/j.1525-1594.2011.01215.x. PMID 21401663
- [Background] Kesar TM, Perumal R, Reisman DS, Jancosko A, Rudolph KS, Higginson JS, Binder-Macleod SA. Functional electrical stimulation of ankle plantarflexor and dorsiflexor muscles: effects on poststroke gait. Stroke. 2009 Dec;40(12):3821-7. doi: 10.1161/STROKEAHA.109.560375. Epub 2009 Oct 15. PMID 19834018
- [Background] Awad LN, Reisman DS, Kesar TM, Binder-Macleod SA. Targeting paretic propulsion to improve poststroke walking function: a preliminary study. Arch Phys Med Rehabil. 2014 May;95(5):840-8. doi: 10.1016/j.apmr.2013.12.012. Epub 2013 Dec 28. PMID 24378803
- [Background] Nadeau S, Gravel D, Arsenault AB, Bourbonnais D. Plantarflexor weakness as a limiting factor of gait speed in stroke subjects and the compensating role of hip flexors. Clin Biomech (Bristol). 1999 Feb;14(2):125-35. doi: 10.1016/s0268-0033(98)00062-x. PMID 10619100
- [Background] Chen G, Patten C, Kothari DH, Zajac FE. Gait differences between individuals with post-stroke hemiparesis and non-disabled controls at matched speeds. Gait Posture. 2005 Aug;22(1):51-6. doi: 10.1016/j.gaitpost.2004.06.009. PMID 15996592
- [Background] Awad LN, Hsiao H, Binder-Macleod SA. Central Drive to the Paretic Ankle Plantarflexors Affects the Relationship Between Propulsion and Walking Speed After Stroke. J Neurol Phys Ther. 2020 Jan;44(1):42-48. doi: 10.1097/NPT.0000000000000299. PMID 31834220
- [Background] Bae J, Siviy C, Rouleau M, Menard N, O'Donnell K, Galiana I, Athanassiu M, Ryan D, Bibeau C, Sloot L, Kudzia P, Ellis T, Awad L, Walsh CJ. A lightweight and efficient portable soft exosuit for particular ankle assistance in walking after stroke. IEEE International Conference on Robotics and Automation (ICRA). 2018; 2820-2827.
- [Background] Bowden MG, Balasubramanian CK, Neptune RR, Kautz SA. Anterior-posterior ground reaction forces as a measure of paretic leg contribution in hemiparetic walking. Stroke. 2006 Mar;37(3):872-6. doi: 10.1161/01.STR.0000204063.75779.8d. Epub 2006 Feb 2. PMID 16456121
- [Background] Roelker SA, Bowden MG, Kautz SA, Neptune RR. Paretic propulsion as a measure of walking performance and functional motor recovery post-stroke: A review. Gait Posture. 2019 Feb;68:6-14. doi: 10.1016/j.gaitpost.2018.10.027. Epub 2018 Oct 25. PMID 30408710
- [Result] Choe DK, Aiello AJ, Spangler JE, Walsh CJ, Awad LN. A Propulsion Neuroprosthesis Improves Overground Walking in Community-Dwelling Individuals After Stroke. IEEE Open J Eng Med Biol. 2024 Jul 4;5:563-572. doi: 10.1109/OJEMB.2024.3416028. eCollection 2024. PMID 39157060
- See also: Results Reference — https://ieeexplore.ieee.org/document/10586842

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic (> 6 months) stroke were screened from a participant pool known to the Boston University Neuromotor Recovery Laboratory. Of the 18 participants screened, 13 participants were eligible for enrollment, and 10 participants completed the study. Exclusions: pacemaker (1), live far away / unwilling to travel (1), joint replacement (1), ankle dorsiflexion less than neutral (2), unable to be contacted (1), medical complications preventing participation (1), not interested (1).
Groups:
- Neuroprosthesis-Assisted Walking Evaluation: Participants with chronic stroke will perform a series of short overground walking evaluations at a self-selected fast walking speed with the neuroprosthesis powered and unpowered. When the neuroprosthesis is powered, it provides active neurostimulation assistance for foot clearance and propulsion. When the neuroprosthesis is unpowered, it is worn by the participant but does not provide active assistance.
  The propulsion neuroprosthesis is a textile-based neurostimulation system worn on the waist and paretic lower limb that delivers neurostimulation assistance via electroconductive pads placed on the skin over the target muscles. The neuroprosthesis provides dorsiflexor stimulation during swing phase for foot clearance and plantarflexor stimulation during stance phase for propulsion, delivered synchronously based on integrated sensors detecting the wearer's gait pattern.
Period: Overall Study
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
  Other | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 0
  Race: Black or African American | 0
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: White | 6
  Race: More than one race | 0
  Race: Unknown or Not Reported | 2
  Race: Other: Iranian | 1
  Race: Other: Puerto Rican | 1
Paretic Side [Count of Participants; unit: Participants] — Side of body most affected by the stroke.
  Participants
    Left | 6
    Right | 4
Stroke Chronicity [Mean (Standard Deviation); unit: years] — Length of time since onset of stroke, assessed at study start.
  years | 7.5 (4.5)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 176 (9)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 87.77 (19.68)
Comfortable Walking Speed [Mean (Standard Deviation); unit: meters per second (m/s)] — Speed of self-selected comfortable walking pace measured during the 10-Meter Walk Test (10mWT), a clinical assessment of walking speed.
  meters per second (m/s) | 0.93 (0.23)
Fast Walking Speed [Mean (Standard Deviation); unit: meters per second (m/s)] — Speed of self-selected fast walking pace measured during the 10-Meter Walk Test (10mWT), a clinical assessment of walking speed.
  meters per second (m/s) | 1.24 (0.42)
Paretic Propulsion [Mean (Standard Deviation); unit: percent bodyweight (%bw)] — Peak anterior-posterior ground reaction force of the paretic limb, measured at a self-selected comfortable pace during the 10-Meter Walk Test.
  percent bodyweight (%bw) | 8.50 (4.60)
Propulsion Symmetry [Mean (Standard Deviation); unit: percent (%)] — The contribution of the paretic limb to the total propulsion impulse (i.e., propulsion impulse of the paretic limb divided by the total propulsion impulse, paretic + nonparetic), measured at a self-selected comfortable pace during the 10-Meter Walk Test. Propulsion impulse is the area under the positive portion of the anterior-posterior ground reaction force curve.
  percent (%) | 28.4 (12.2)
Dorsiflexion Angle [Mean (Standard Deviation); unit: degrees] — Peak ankle angle during swing phase, measured at a self-selected comfortable pace during the 10-Meter Walk Test.
  degrees | 2.07 (5.04)
Dorsiflexor Impairment [Count of Participants; unit: Participants] — Number of participants with paretic dorsiflexion angle during swing phase that is less than neutral (90-degree angle between foot and shank).
  Participants
    Dorsiflexor Impairment | 3
    No Dorsiflexor Impairment | 7

OUTCOME MEASURES:

1. Primary Outcome: Immediate Change in Walking Speed
Description: Change in walking speed from unassisted walking to walking with neurostimulation assistance at either an early or a late timing, measured at a self-selected fast pace across a straight 10-meter walkway. Early timing of plantarflexor neurostimulation was delivered at 40% of paretic limb support phase (before mid-stance). Late timing of plantarflexor neurostimulation was delivered at 60% of paretic limb support phase (after mid-stance).
Time Frame: Early Neurostimulation Timing Condition (40% stance); Late Neurostimulation Timing Condition (60% stance)
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
meters per second (m/s)
  Early Neurostimulation Timing (40% stance) | 0.01 (0.01)
  Late Neurostimulation Timing (60% stance) | 0.03 (0.02)

2. Primary Outcome: Immediate Change in Paretic Propulsion
Description: Change in paretic propulsion from unassisted walking to walking with neurostimulation assistance at either an early or a late timing, measured at a self-selected fast pace across a straight 10-meter walkway. Early timing of plantarflexor neurostimulation was delivered at 40% of paretic limb support phase (before mid-stance). Late timing of plantarflexor neurostimulation was delivered at 60% of paretic limb support phase (after mid-stance). Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Time Frame: Early Neurostimulation Timing Condition (40% stance); Late Neurostimulation Timing Condition (60% stance)
Measure: Mean (Standard Error); unit: percent bodyweight (%bw)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent bodyweight (%bw)
  Early Neurostimulation Timing Condition (40% stance) | 0.35 (0.41)
  Late Neurostimulation Timing Condition (60% stance) | 0.71 (0.60)

3. Primary Outcome: Immediate Change in Propulsion Symmetry
Description: Change in propulsion symmetry from unassisted walking to walking with neurostimulation assistance at either an early or a late timing, measured at a self-selected fast pace across a straight 10-meter walkway. Early timing of plantarflexor neurostimulation was delivered at 40% of paretic limb support phase (before mid-stance). Late timing of plantarflexor neurostimulation was delivered at 60% of paretic limb support phase (after mid-stance). Propulsion symmetry was calculated as the propulsion impulse of the paretic limb divided by the total propulsion impulse (paretic + nonparetic). Propulsion impulse is the area under the positive portion of the anterior-posterior ground reaction force curve.
Time Frame: Early Neurostimulation Timing Condition (40% stance); Late Neurostimulation Timing Condition (60% stance)
Measure: Mean (Standard Error); unit: percent (%)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent (%)
  Early Neurostimulation Timing Condition (40% stance) | -0.02 (1.19)
  Late Neurostimulation Timing Condition (60% stance) | -0.92 (1.16)

4. Primary Outcome: Immediate Change in Walking Speed
Description: Change in walking speed from unassisted walking to walking with neurostimulation assistance at either an early timing or an individual-specific preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Early timing of plantarflexor neurostimulation was delivered at 40% of paretic limb support phase (before mid-stance). Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion.
Time Frame: Early Neurostimulation Timing Condition (40% stance); Preferred Neurostimulation Timing Condition (propulsion-based tuning)
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
meters per second (m/s)
  Early Neurostimulation Timing Condition (40% stance) | 0.01 (0.01)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 0.03 (0.01)

5. Primary Outcome: Immediate Change in Paretic Propulsion
Description: Change in paretic propulsion from unassisted walking to walking with neurostimulation assistance at either an early timing or an individual-specific preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Early timing of plantarflexor neurostimulation was delivered at 40% of paretic limb support phase (before mid-stance). Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Time Frame: as for outcome 4
Measure: Mean (Standard Error); unit: percent bodyweight (%bw)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent bodyweight (%bw)
  Early Neurostimulation Timing Condition (40% stance) | 0.35 (0.41)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 1.41 (0.48)

6. Primary Outcome: Immediate Change in Propulsion Symmetry
Description: Change in propulsion symmetry from unassisted walking to walking with neurostimulation assistance at either an early timing or an individual-specific preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Early timing of plantarflexor neurostimulation was delivered at 40% of paretic limb support phase (before mid-stance). Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Propulsion symmetry was calculated as the propulsion impulse of the paretic limb divided by the total propulsion impulse (paretic + nonparetic). Propulsion impulse is the area under the positive portion of the anterior-posterior ground reaction force curve.
Time Frame: as for outcome 4
Measure: Mean (Standard Error); unit: percent (%)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent (%)
  Early Neurostimulation Timing Condition (40% stance) | -0.02 (1.19)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 1.19 (1.26)

7. Primary Outcome: Immediate Change in Walking Speed
Description: Change in walking speed from unassisted walking to walking with neurostimulation assistance at either a late timing or an individual-specific preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Late timing of plantarflexor neurostimulation was delivered at 60% of paretic limb support phase (before mid-stance). Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion.
Time Frame: Late Neurostimulation Timing Condition (60% stance); Preferred Neurostimulation Timing Condition (propulsion-based tuning)
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
meters per second (m/s)
  Late Neurostimulation Timing Condition (60% stance) | 0.03 (0.02)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 0.03 (0.01)

8. Primary Outcome: Immediate Change in Paretic Propulsion
Description: Change in paretic propulsion from unassisted walking to walking with neurostimulation assistance at either a late timing or an individual-specific preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Late timing of plantarflexor neurostimulation was delivered at 60% of paretic limb support phase (after mid-stance). Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Time Frame: as for outcome 7
Measure: Mean (Standard Error); unit: percent bodyweight (%bw)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent bodyweight (%bw)
  Late Neurostimulation Timing Condition (60% stance) | 0.71 (0.60)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 1.41 (0.48)

9. Primary Outcome: Immediate Change in Propulsion Symmetry
Description: Change in propulsion symmetry from unassisted walking to walking with neurostimulation assistance at either a late timing or an individual-specific preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Late timing of plantarflexor neurostimulation was delivered at 60% of paretic limb support phase (before mid-stance). Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Propulsion symmetry was calculated as the propulsion impulse of the paretic limb divided by the total propulsion impulse (paretic + nonparetic). Propulsion impulse is the area under the positive portion of the anterior-posterior ground reaction force curve.
Time Frame: as for outcome 7
Measure: Mean (Standard Error); unit: percent (%)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent (%)
  Late Neurostimulation Timing Condition (60% stance) | -0.92 (1.16)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 1.19 (1.26)

10. Primary Outcome: Immediate Change in Walking Speed
Description: Change in walking speed from unassisted walking to walking with neurostimulation assistance at either a non-preferred or a preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion.
Time Frame: Non-Preferred Neurostimulation Timing Condition (propulsion-based tuning); Preferred Neurostimulation Timing Condition (propulsion-based tuning)
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
meters per second (m/s)
  Non-Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 0.00 (0.02)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 0.03 (0.01)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; An a priori power analysis (G*Power 3.1.9.7) determined that a sample size of 10 participants could detect an effect size (Cohen's D) of 1.0 with 80% power and alpha = 0.05; Test type: Other — Single group test of difference; p = 0.131, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.525; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.01 to 0.07], Standard Error of Mean 0.02 — Difference = Preferred Timing - Non-Preferred Timing

11. Primary Outcome: Immediate Change in Paretic Propulsion
Description: Change in paretic propulsion from unassisted walking to walking with neurostimulation assistance at either a non-preferred or a preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Time Frame: as for outcome 10
Measure: Mean (Standard Error); unit: percent bodyweight (%bw)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent bodyweight (%bw)
  Non-Preferred Neurostimulation Timing Condition (propulsion-based tuning) | -0.36 (0.36)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 1.41 (0.48)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.001, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 1.623; Mean Difference (Final Values) = 1.77, 95% CI 2-sided [0.99 to 2.56], Standard Error of Mean 0.35 — Difference = Preferred Timing - Non-Preferred Timing

12. Primary Outcome: Immediate Change in Propulsion Symmetry
Description: Change in propulsion symmetry from unassisted walking to walking with neurostimulation assistance at either a non-preferred or a preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Propulsion symmetry was calculated as the propulsion impulse of the paretic limb divided by the total propulsion impulse (paretic + nonparetic). Propulsion impulse is the area under the positive portion of the anterior-posterior ground reaction force curve.
Time Frame: as for outcome 10
Measure: Mean (Standard Error); unit: percent (%)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent (%)
  Non-Preferred Neurostimulation Timing Condition (propulsion-based tuning) | -2.13 (0.78)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 1.19 (1.26)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.017, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.923; Mean Difference (Final Values) = 3.32, 95% CI 2-sided [0.75 to 5.89], Standard Error of Mean 1.14 — Difference = Preferred Timing - Non-Preferred Timing

13. Primary Outcome: Walking Speed at Non-Preferred Timing
Description: Walking speed with or without neurostimulation assistance measured at a self-selected fast pace across a straight 10-meter walkway.
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
meters per second (m/s)
  Unassisted Walking Condition | 1.30 (0.14)
  Assisted Walking Condition | 1.30 (0.15)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.874, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.052; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.034 to 0.039], Standard Error of Mean 0.016 — Difference = Assisted - Unassisted

14. Primary Outcome: Paretic Propulsion at Non-Preferred Timing
Description: Paretic propulsion with or without neurostimulation assistance measured at a self-selected fast pace across a straight 10-meter walkway. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: percent bodyweight (%bw)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent bodyweight (%bw)
  Unassisted Walking Condition | 12.19 (1.51)
  Assisted Walking Condition | 11.83 (1.73)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.345, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = -0.315; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.18 to 0.46], Standard Error of Mean 0.36 — Difference = Assisted - Unassisted

15. Primary Outcome: Propulsion Symmetry at Non-Preferred Timing
Description: Propulsion symmetry with or without neurostimulation assistance measured at a self-selected fast pace across a straight 10-meter walkway. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb. Propulsion symmetry was calculated as the propulsion impulse of the paretic limb divided by the total propulsion impulse (paretic + nonparetic). Propulsion impulse is the area under the positive portion of the anterior-posterior ground reaction force curve.
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: percent (%)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent (%)
  Unassisted Walking Condition | 32.2 (2.7)
  Assisted Walking Condition | 30.0 (3.1)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.024, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = -0.859; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-3.90 to -0.36], Standard Error of Mean 0.78 — Difference = Assisted - Unassisted

16. Primary Outcome: Walking Speed at Preferred Timing
Description: as for outcome 13
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
meters per second (m/s)
  Unassisted Walking Condition | 1.31 (0.15)
  Assisted Walking Condition | 1.34 (0.15)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.044, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.739; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [0.00 to 0.06], Standard Error of Mean 0.01 — Difference = Assisted - Unassisted

17. Primary Outcome: Paretic Propulsion at Preferred Timing
Description: as for outcome 14
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: percent bodyweight (%bw)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent bodyweight (%bw)
  Unassisted Walking Condition | 11.87 (1.71)
  Assisted Walking Condition | 13.28 (1.89)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.017, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.928; Mean Difference (Final Values) = 1.41, 95% CI 2-sided [0.32 to 2.50], Standard Error of Mean 0.48 — Difference = Assisted - Unassisted

18. Primary Outcome: Propulsion Symmetry at Preferred Timing
Description: as for outcome 15
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: percent (%)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent (%)
  Unassisted Walking Condition | 31.8 (3.1)
  Assisted Walking Condition | 33.0 (3.4)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.372, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.297; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-1.67 to 4.04], Standard Error of Mean 1.26 — Difference = Assisted - Unassisted

19. Primary Outcome: Unassisted Fast Walking Speed
Description: Walking speed without neurostimulation assistance measured at a self-selected fast pace using the 10-Meter Walk Test.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
meters per second (m/s)
  Pre-Intervention | 1.24 (0.13)
  Post-Intervention | 1.38 (0.14)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.001, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 1.508; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [0.07 to 0.20], Standard Error of Mean 0.03 — Difference = Post-Session - Pre-Session

20. Primary Outcome: Unassisted Paretic Propulsion at Fast Speed
Description: Paretic propulsion during walking without neurostimulation assistance at a self-selected fast pace during the 10-Meter Walk Test. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: percent bodyweight (%bw)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent bodyweight (%bw)
  Pre-Intervention | 11.20 (1.91)
  Post-Intervention | 13.44 (1.53)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.043, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.746; Mean Difference (Final Values) = 2.24, 95% CI 2-sided [0.09 to 4.39], Standard Error of Mean 0.95 — Difference = Post-Session - Pre-Session

21. Primary Outcome: Unassisted Propulsion Symmetry at Fast Speed
Description: Propulsion symmetry during walking without neurostimulation assistance at a self-selected fast pace during the 10-Meter Walk Test. Propulsion symmetry was calculated as the propulsion impulse of the paretic limb divided by the total propulsion impulse (paretic + nonparetic). Propulsion impulse is the area under the positive portion of the anterior-posterior ground reaction force curve.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: percent (%)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent (%)
  Pre-Intervention | 28.7 (4.0)
  Post-Intervention | 33.2 (3.2)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.041, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.752; Mean Difference (Final Values) = 4.53, 95% CI 2-sided [0.22 to 8.83], Standard Error of Mean 1.90 — Difference = Post-Session - Pre-Session

22. Primary Outcome: Unassisted Comfortable Walking Speed
Description: Walking speed without neurostimulation assistance measured at a self-selected comfortable pace using the 10-Meter Walk Test.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: meters per second (m/s)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
meters per second (m/s)
  Pre-Intervention | 0.93 (0.07)
  Post-Intervention | 1.06 (0.08)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.013, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.983; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.03 to 0.21], Standard Error of Mean 0.04 — Difference = Post-Session - Pre-Session

23. Primary Outcome: Unassisted Paretic Propulsion at Comfortable Speed
Description: Paretic propulsion during walking without neurostimulation assistance at a self-selected comfortable pace during the 10-Meter Walk Test. Paretic propulsion was calculated as the peak anterior-posterior ground reaction force of the paretic limb.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: percent bodyweight (%bw)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent bodyweight (%bw)
  Pre-Intervention | 8.50 (1.46)
  Post-Intervention | 10.12 (1.24)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.012, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.985; Mean Difference (Final Values) = 1.61, 95% CI 2-sided [0.44 to 2.78], Standard Error of Mean 0.52 — Difference = Post-Session - Pre-Session

24. Primary Outcome: Unassisted Propulsion Symmetry at Comfortable Speed
Description: Propulsion symmetry during walking without neurostimulation assistance at a self-selected comfortable pace during the 10-Meter Walk Test. Propulsion symmetry was calculated as the propulsion impulse of the paretic limb divided by the total propulsion impulse (paretic + nonparetic). Propulsion impulse is the area under the positive portion of the anterior-posterior ground reaction force curve.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: percent (%)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
percent (%)
  Pre-Intervention | 28.4 (3.9)
  Post-Intervention | 33.2 (3.4)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.036, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.779; Mean Difference (Final Values) = 4.75, 95% CI 2-sided [0.39 to 9.11], Standard Error of Mean 1.93 — Difference = Post-Session - Pre-Session

25. Secondary Outcome: Onset Timing of Plantarflexor Neurostimulation
Description: The timepoint in the gait cycle when plantarflexor neurostimulation turns on. Early timing of plantarflexor neurostimulation was set at 40% of paretic limb support phase (before mid-stance). Late timing of plantarflexor neurostimulation was set at 60% of paretic limb support phase (after mid-stance). Actual delivery of neurostimulation may vary based on the inertial sensor based real-time control and sensing of gait features.
Time Frame: Early Neurostimulation Timing Condition (40% stance); Late Neurostimulation Timing Condition (60% stance)
Population: Neurostimulation timing information was not available for 2 participants due to issues with data streaming from the neuroprosthesis.
Measure: Mean (Standard Deviation); unit: percent stance (% stance)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 8
percent stance (% stance)
  Early Neurostimulation Timing Condition (40% stance) | 46.9 (2.0)
  Late Neurostimulation Timing Condition (60% stance) | 63.7 (2.0)

26. Secondary Outcome: Preferred Neurostimulation Timing
Description: Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Early timing of plantarflexor neurostimulation was delivered at 40% of paretic limb support phase (before mid-stance). Late timing of plantarflexor neurostimulation was delivered at 60% of paretic limb support phase (after mid-stance).
Time Frame: Preferred Neurostimulation Timing Condition (propulsion-based tuning)
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
Participants
  Early Neurostimulation Timing Condition (40% stance) | 5
  Late Neurostimulation Timing Condition (60% stance) | 5

27. Secondary Outcome: Dorsiflexion Angle (No Dorsiflexor Impairment)
Description: Dorsiflexion angle during walking at a self-selected fast pace across a straight 10-meter walkway for the subset of participants without paretic dorsiflexor impairment. Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Dorsiflexion angle is the positive angle between the foot and the shank from a neutral 90-degree position, measured using optical motion capture.
Time Frame: Pre-Intervention; Non-Preferred Neurostimulation Timing Condition (propulsion-based tuning); Preferred Neurostimulation Timing Condition (propulsion-based tuning)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 7
degrees
  Pre-Intervention | 4.50 (3.56)
  Non-Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 5.15 (5.52)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 5.14 (5.25)

28. Secondary Outcome: Dorsiflexion Angle (With Dorsiflexor Impairment)
Description: Dorsiflexion angle during walking at a self-selected fast pace across a straight 10-meter walkway for the subset of participants with paretic dorsiflexor impairment. Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Dorsiflexion angle is the positive angle between the foot and the shank from a neutral 90-degree position, measured using optical motion capture. Negative dorsiflexion angle indicates plantarflexion of the foot, downwards from a neutral 90-degree position.
Time Frame: as for outcome 27
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 3
degrees
  Pre-Intervention | -3.61 (2.70)
  Non-Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 0.13 (4.22)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | -1.03 (3.40)

29. Secondary Outcome: Immediate Change in Dorsiflexion Angle
Description: Change in dorsiflexion angle from unassisted walking to walking with neurostimulation assistance at either a non-preferred or a preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Dorsiflexion angle is the positive angle between the foot and the shank from a neutral 90-degree position, measured using optical motion capture.
Time Frame: as for outcome 10
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
degrees
  Non-Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 1.48 (0.95)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 1.46 (0.94)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.962, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = -0.015; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-1.24 to 1.19], Standard Error of Mean 0.54 — Difference = Preferred Timing - Non-Preferred Timing

30. Secondary Outcome: Immediate Change in Plantarflexor Power
Description: Change in plantarflexor power from unassisted walking to walking with neurostimulation assistance at either a non-preferred or a preferred timing, measured at a self-selected fast pace across a straight 10-meter walkway. Timing preference was determined for each participant individually based on which of the early or late timings produced greater paretic propulsion. Plantarflexor power is the peak rate of change in the rotation force of the foot towards the ground, measured using optical motion capture.
Time Frame: as for outcome 10
Measure: Mean (Standard Error); unit: watt per kilogram (W/kg)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
watt per kilogram (W/kg)
  Non-Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 0.13 (0.08)
  Preferred Neurostimulation Timing Condition (propulsion-based tuning) | 0.27 (0.07)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.146, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.504; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.06 to 0.35], Standard Error of Mean 0.09 — Difference = Preferred Timing - Non-Preferred Timing

31. Secondary Outcome: Dorsiflexion Angle at Non-Preferred Timing
Description: Dorsiflexion angle with or without neurostimulation assistance measured at a self-selected fast pace across a straight 10-meter walkway. Dorsiflexion angle is the positive angle between the foot and the shank from a neutral 90-degree position, measured using optical motion capture.
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
degrees
  Unassisted Walking Condition | 2.16 (1.93)
  Assisted Walking Condition | 3.64 (1.74)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.152, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.495; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [-0.66 to 3.63], Standard Error of Mean 0.95 — Difference = Assisted - Unassisted

32. Secondary Outcome: Plantarflexor Power at Non-Preferred Timing
Description: Plantarflexor power with or without neurostimulation assistance measured at a self-selected fast pace across a straight 10-meter walkway. Plantarflexor power is the peak rate of change in the rotation force of the foot towards the ground, measured using optical motion capture.
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: watts per kilogram (W/kg)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
watts per kilogram (W/kg)
  Unassisted Walking Condition | 1.88 (0.17)
  Assisted Walking Condition | 2.00 (0.20)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.153, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.494; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.06 to 0.31], Standard Error of Mean 0.08 — Difference = Assisted - Unassisted

33. Secondary Outcome: Dorsiflexion Angle at Preferred Timing
Description: as for outcome 31
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
degrees
  Unassisted Walking Condition | 1.83 (1.98)
  Assisted Walking Condition | 3.29 (1.73)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.155, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.491; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [-0.67 to 3.58], Standard Error of Mean 0.94 — Difference = Assisted - Unassisted

34. Secondary Outcome: Plantarflexor Power at Preferred Timing
Description: as for outcome 32
Time Frame: Unassisted Walking Condition; Assisted Walking Condition
Measure: Mean (Standard Error); unit: watts per kilogram (W/kg)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
watts per kilogram (W/kg)
  Unassisted Walking Condition | 1.84 (0.20)
  Assisted Walking Condition | 2.11 (0.21)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.004, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 1.199; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [0.11 to 0.43], Standard Error of Mean 0.07 — Difference = Assisted - Unassisted

35. Secondary Outcome: Unassisted Dorsiflexion Angle at Fast Speed
Description: Dorsiflexion angle during walking without neurostimulation assistance at a self-selected fast pace during the 10-Meter Walk Test. Dorsiflexion angle is the positive angle between the foot and the shank from a neutral 90-degree position, measured using optical motion capture.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
degrees
  Pre-Intervention | 2.85 (1.98)
  Post-Intervention | 0.66 (1.65)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.014, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = -0.962; Mean Difference (Final Values) = -2.19, 95% CI 2-sided [-3.82 to -0.56], Standard Error of Mean 0.72 — Difference = Post-Session - Pre-Session

36. Secondary Outcome: Unassisted Plantarflexor Power at Fast Speed
Description: Plantarflexor power during walking without neurostimulation assistance at a self-selected fast pace during the 10-Meter Walk Test. Plantarflexor power is the peak rate of change in the rotation force of the foot towards the ground, measured using optical motion capture.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: watt per kilogram (W/kg)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
watt per kilogram (W/kg)
  Pre-Intervention | 1.78 (0.20)
  Post-Intervention | 1.98 (0.20)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.350, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.312; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.26 to 0.66], Standard Error of Mean 0.20 — Difference = Post-Session - Pre-Session

37. Secondary Outcome: Unassisted Dorsiflexion Angle at Comfortable Speed
Description: Dorsiflexion angle during walking without neurostimulation assistance at a self-selected comfortable pace during the 10-Meter Walk Test. Dorsiflexion angle is the positive angle between the foot and the shank from a neutral 90-degree position, measured using optical motion capture.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
degrees
  Pre-Intervention | 2.07 (1.59)
  Post-Intervention | 0.27 (1.82)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.052, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = -0.706; Mean Difference (Final Values) = -1.80, 95% CI 2-sided [-3.63 to 0.02], Standard Error of Mean 0.81 — Difference = Post-Session - Pre-Session

38. Secondary Outcome: Unassisted Plantarflexor Power at Comfortable Speed
Description: Plantarflexor power during walking without neurostimulation assistance at a self-selected comfortable pace during the 10-Meter Walk Test. Plantarflexor power is the peak rate of change in the rotation force of the foot towards the ground, measured using optical motion capture.
Time Frame: Pre-Intervention; Post-Intervention
Measure: Mean (Standard Error); unit: watt per kilogram (W/kg)
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
Number analyzed (Participants) | 10
watt per kilogram (W/kg)
  Pre-Intervention | 1.25 (0.12)
  Post-Intervention | 1.39 (0.07)
Statistical Analysis 1: Comparison: Neuroprosthesis-Assisted Walking Evaluation; [analysis description as in outcome 10, analysis 1]; Test type: Other — Single group test of difference; p = 0.221, t-test, 2 sided — alpha = 0.05; Effect Size (Cohen's D) = 0.416; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.10 to 0.39], Standard Error of Mean 0.11 — Difference = Post-Session - Pre-Session

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Neuroprosthesis-Assisted Walking Evaluation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Data streaming issue led to two participants not having information about the timing of neurostimulation assistance during the gait cycle.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT06459401/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT06459401/SAP_001.pdf